CLINICAL TRIAL: NCT01694459
Title: Comparison of Low-dose Heparin Versus Standard Dose Heparin During Coronary Interventions (DEDICA Trial)
Brief Title: DEDICA (Dose of HEparin During Coronary Angioplasty) Trial
Acronym: DEDICA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Filippo Neri General Hospital (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Vincenzo Pasceri, Attending Cardiologist, San Filippo Neri General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 596-2012-D
Record Dates: First submitted 2012-09-23; First posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Stable Angina; Angina, Unstable; Non-ST Elevation (NSTEMI) Myocardial Infarction
Keywords: angioplasty; heparin; trial
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction; Myocardial Infarction | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dose heparin (Active Comparator): Bolus of 100 UI/Kg of heparin. Activated clotting time (ACT) > 300 sec. during the procedure
  Interventions: Drug: Standard dose heparin
- Low-dose heparin (Experimental): Bolus of 50 UI/Kg heparin with a target ACT during the procedure of >200 sec.
  Interventions: Drug: Low-dose heparin

INTERVENTIONS:
Drug: Low-dose heparin — Bolus of 50 UI/Kg of heparin at the beginning of coronary interventions
  Other Names: 50 UI/Kg bolus heparin
  Arms: Low-dose heparin
Drug: Standard dose heparin — Bolus of 100 UI/Kg of heparin at the beginning of coronary interventional procedure.
  Other Names: 100 Ui/Kg bolus heparin
  Arms: Standard dose heparin

SUMMARY:
International guidelines support the use of a full-dose heparin (anticoagulants) during coronary intervention. However, a lower dose of heparin may be adequate, thanks to advances in angioplasty techniques and the widespread use of pretreatment with two antiplatelet agents.

Thus the investigators designed a study comparing safety and efficacy of standard dose heparin (100 UI/Kg) versus low-dose (50 UI/Kg) in patients undergoing coronary angioplasty who are on aspirin and clopidogrel at the time of the procedure.

DETAILED DESCRIPTION:
* Patients undergoing coronary angioplasty will be randomised to standard vs. low-dose heparin. the study will include "all-comers" (patients with either stable angina or acute coronary syndromes); only patients with ST-elevation myocardial infarction will be excluded.
* An ACT (activated clotting time) will be performed after the initial bolus of heparin: for the standard dose group the target ACT will be > 300 sec. (as recommended by guidelines) while for the low-dose the target ACT will be > 180 sec.

Aim of the study is to show equivalence in ischemic events between the two doses of heparin, in order to confirm the safety of lower dose of heparin in contemporary coronary interventions.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina, unstable angina or Non-ST elevation myocardial infarction undergoing coronary angioplasty.
* Mandatory pretreatment with aspirin and clopidogrel

Exclusion Criteria:

* ST elevation myocardial infarction
* Coronary interventions with rotational atherectomy
* Coronary interventions on chronic total occlusions (CTO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
MACE + stent thrombosis + major bleeding (TIMI definition) | 30 days
  MACE (death, myocardial infarction, target vessel revascularization) + stent thrombosis + major bleeding (TIMI definition)

SECONDARY OUTCOMES:
MACE | 30 days
  MACE = death, myocardial infarction, target vessel revascularization
Major Bleeding | 30 days
  Major bleeding according to TIMI criteria
Stent thrombosis | 30 days
  Stent thrombosis (definite or probable according to ARC criteria)
CK-MB increase | 30 days
  Any CK MB increase >3 times upper limit of normal or >50% baseline levels (if baseline levels already >then upper limit of normal)

OTHER OUTCOMES:
Major bleeding | 30 days
  Major bleeding according to STEEPLE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Pasceri, MD, Study Chair — San Filippo Neri Hospital; Francesco Pelliccia, MD, Study Director — University of Roma La Sapienza
Locations (1):
- University of Rome La Sapienza, Rome, Italy